CLINICAL TRIAL: NCT06240780
Title: A Randomized Prospective Study to Evaluate the Incrediwear Products Immediately After ACL or ACL+MCL Arthroscopic Surgery
Brief Title: Incrediwear ACL MCL Arthroscopic Surgery Recovery Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma Joint Reconstruction Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-04
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Arthroscopic Surgical Procedures; Anterior Cruciate Ligament Reconstruction
Keywords: Arthroscopic Surgical Procedures; Anterior Cruciate Ligament Reconstruction; Medial Collateral Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: . Participants will randomly be assigned treatment type in addition to the standard of care procedure they will be instructed to follow (active vs. placebo vs standard of care alone) based on surgery type. An equal number of patients from each primary condition type (ACL or ACL+MCL) will be assigned to each treatment type.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded stratified randomization of subjects from two arms into one of three groups per arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ACL Arthroscopic Active Participants (Active Comparator): After the surgery, the patient will be placed in the study provided semiconductor element interwoven Incrediwear Leg Sleeve from the ankle to the thigh and the Incrediwear sock, on the operative leg, and a thigh high compression hose on the non operative leg, worn 23 hours per day. At day 31 patient will wear the leg sleeve at night and be placed in the Incrediwear Knee Sleeve.
  Interventions: Other: Activated Incrediwear Products
- ACL Arthroscopic Placebo Participants (Placebo Comparator): After the surgery, the patient will be placed in the study provided plain fabric Incrediwear Leg Sleeve from the ankle to the thigh and the Incrediwear sock, on the operative leg, and a thigh high compression hose on the non operative leg, worn 23 hours per day. At day 31 patient will wear the leg sleeve at night and be placed in the Incrediwear Knee Sleeve.
  Interventions: Other: Sham Incrediwear Products
- ACL Arthroscopic Stand of Care Participants (No Intervention): After the surgery, the patient will be placed in thigh high compression hose, bilaterally, worn 23 hours per day for 31 days.
- ACL + MCL Arthroscopic Active Participants (Active Comparator): After the surgery, the patient will be placed in the study provided semiconductor element interwoven Incrediwear Leg Sleeve from the ankle to the thigh and the Incrediwear sock, on the operative leg, and a thigh high compression hose on the non operative leg, worn 23 hours per day. At day 31 patient will wear the leg sleeve at night and be placed in the Incrediwear Knee Sleeve.
  Interventions: Other: Activated Incrediwear Products
- ACL + MCL Arthroscopic Placebo Participants (Placebo Comparator): After the surgery, the patient will be placed in the study provided plain fabric Incrediwear Leg Sleeve from the ankle to the thigh and the Incrediwear sock, on the operative leg, and a thigh high compression hose on the non operative leg, worn 23 hours per day. At day 31 patient will wear the leg sleeve at night and be placed in the Incrediwear Knee Sleeve.
  Interventions: Other: Sham Incrediwear Products
- ACL + MCL Arthroscopic Stand of Care Participants (No Intervention): After the surgery, the patient will be placed in thigh high compression hose, bilaterally, worn 23 hours per day for 31 days.

INTERVENTIONS:
Other: Activated Incrediwear Products — Activated Incrediwear products incorporates semiconductor elements within the fabric that releases negative ions when stimulated by body heat. The negative ions activate cellular vibrations that increase blood flow and circulation.
  Arms: ACL + MCL Arthroscopic Active Participants; ACL Arthroscopic Active Participants
Other: Sham Incrediwear Products — Simple fabric Incrediwear products that do not include the semiconductor elements within the fabric.
  Arms: ACL + MCL Arthroscopic Placebo Participants; ACL Arthroscopic Placebo Participants

SUMMARY:
The goal of this clinical trial is to assess the benefits of using the Incrediwear knee products after anterior cruciate ligament arthroscopic surgery or anterior cruciate ligament and medial collateral ligament (ACL+MCL) arthroscopic surgery, on the postoperative pain, range of motion and effusion. Participant population includes female or male patients in relative good health, 18 to 65 years old. The investigators will compare participants with Incrediwear and placebo Incrediwear products during the first 6-month postoperative period. The main question it aims to answer are:

* Will the Incrediwear products help participants to decrease postoperative pain and swelling?
* Will the Incrediwear products help the participants by increasing the range of motion in a shorter amount of time than the placebo group? Participants will be asked to maintain a journal documenting surgical site pain, pain medication type and quantity taken.

Researcher will compare 90 participants enrolled in one of six groups, double blinded and randomly assigned, to see if the Incrediwear products assist in controlling postoperative swelling, and increase range of motion in a shorter amount of time.

* ACL participants randomly assigned the Incrediwear product, placebo product, or none
* ACL+MCL participants randomly assigned the Incrediwear product, placebo product, or none

DETAILED DESCRIPTION:
Researcher will identify patients of the Primary Investigator (PI) who are candidate for the study. Subjects must otherwise be in good health as determined by medical history, physical examination, vital signs, and applicable laboratory tests and receive medical clearance for the procedure by the PI.

Subjects must be able to read and sign an informed consent form indicating understand the purpose of, and the procedures required for the study, and are willing to participate and comply with the study protocol.

This will be a prospective study to evaluate the benefit of the Incrediwear product after ACL repair or ACL+MCL repair via arthroscopic surgery. Subjects who fit the inclusion and exclusion criteria will be reviewed on a subject-by-subject basis at the time of informed consent documentation.

Preoperative and Post-Operative Measurements:

Subjective: Participants rates surgical site pain, on a 0-10 Visual Analogue Scale (VAS) pain scale.

Participants will record pain medication type and quantity taken in a daily pain diary.

Objective: Surgical extremity range of motion, and surgical extremity knee effusion.

Measurements will be taken at; Preop appointment, Postop Day 0, Day 3, Day 7, Day 14, Day 21, Day 30 (1 month), Day 45, Day 60 (2 month), Day 100 (3 month), and Day 180 (6 month).

After the surgery, the participant will be placed in the study provided Incrediwear Leg Sleeve from the ankle to the thigh and the Incrediwear sock. The Participant will wear the products at all times, for a minimum of 23 hours per day, for days 1 through 30.

At day 31, the participant will wear the leg sleeve at night, knee sleeve during the day, and is no longer required to wear the Incrediwear sock, until day 180.

At the 6 month postoperative appointment, the participant will turn in the patient journal.

ELIGIBILITY:
Inclusion Criteria:

* Consented to protocol
* Compliant to protocol
* BMI less than 35
* Undergoing ACL or ACL+MCL within 30 days

Exclusion Criteria:

* Rheumatoid Arthritis
* Poorly controlled diabetes (HgA1c > 7.5)
* Previous blood clots
* BMI greater than 35
* Varicosities on operative leg
* Pain management patient
* Prior knee surgery to the operative / study knee
* Worker's Comp patients
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Patient Pain Experience | 180 days
  The Visual Analogue Scale (VAS), a 0 to 10 scale, with 0 being no pain and 10 being the worst pain will be used to measures pain intensity.
Pain Medication Usage | 180 days
  Patient will document pain medication type and quantity taken in a daily pain diary.
Effusion/swelling Measurements | 180 days
  The Patella sweep test is used to measure effusion. The measured rating is a quantity on a scale of 0 to 3, with 0 rating no fluid-wave while perorming a downward stroke, 1 a large bulge, 2 medial fluid returns to position without performing a downward sweep, and 3 excell of fluid that makes it impossible to stroke the medial fluid away. Measurements will be taken at set times during the postoperative period.
Range of Motion | 180 days
  The patient's range of motion captured at all time points during the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Steinmetz, MD, Principal Investigator — Oklahoma Joint Reconstruction Institute
Locations (1):
- Oklahoma Joint Reconstruction Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the conclusion of the study, and may be used for publication approximately 6 months after study closes.
Access Criteria: Access to study protocol, SAP,ICF, CSR, and analytic code will be available upon request to the PRS.

REFERENCES:
- See also: Current and past research information regarding the Incrediwear products. — https://incrediwear.com/pages/research